CLINICAL TRIAL: NCT05454813
Title: Evaluation of a Wetness Sensing System for Continence Care
Brief Title: Wetness Sensing System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medline Industries (Industry)
Collaborators: Rochester Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MED-2021-DIV82-002
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-08

CONDITIONS: System Validation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All (Other): Each participant will be provided with the FitRight ® System for the duration of the study. The study products will be used to collect real-life measurement data in order to assess the FitRight® System.
  Interventions: Device: Wetness Sensing System Validation

INTERVENTIONS:
Device: Wetness Sensing System Validation — Participants will use the Wetness Sensing System in a simulated setting in the sitting, supine and side position (participants are randomized to either the left or right side position).

SUMMARY:
The investigational product to be evaluated in this study is FitRight® ConnectTM Wetness Sensing System which includes: the FitRight® ConnectTM Pod, the FitRight® ConnectTM App, the FitRight® ConnectTM charger/adapter and the FitRight® ConnectTM Sensing Brief-(Medline Industries, LP) henceforth, referred to as FitRight® System, Pod, App, Charger, Alert Indicator and Brief. The purpose of this study is to validate the FitRight System sensor's ability to detect when an adult brief has absorbed enough liquid (~90-360 milliliters (mL)) normal saline via simulated urinary void to trigger an alert to change the brief.

DETAILED DESCRIPTION:
Each participant will be provided with the FitRight® System for the duration of the study. The study products will be used to collect real-life measurement data in order to assess the FitRight® System. Each participant will be asked to wear at least three briefs so that they are wearing each brief during the simulated voids performed by the site staff. The site staff will perform the simulated void by addition of (90-360 mL normal saline to the brief. The FitRight® System will be assessed for alerts while participants are in the following positions: supine, sitting, and laying on either left or right side. Each participant will be randomized to either the left or right side. Twenty-two of the fifty-six participants will perform rewet testing procedures. The study results will be used to assess the reliability of the device's absorption to trigger an alert

ELIGIBILITY:
Inclusion Criteria:

* Individuals at least18 years of age
* Individual can dress and undress self with no assistance
* Individuals can ambulate without assistance
* Individual can sit unsupported in a chair or on bedside with no assistance
* Individual can lay supine and propel self up with no assistance
* Individual can lie left/right lateral and propel self up with no assistance
* Individuals who have hip dimensions between 32" and 70" (81-178 cm

Exclusion Criteria:

* Individual is sensitive to the components of the study product(s).
* Individual is considered inappropriate by the Principal Investigator (PI).
* Individual has self-reported current skin condition(s) or issues around the sacral or perineal areas, such as open sores, sacral pressure injuries, rash, burns, surgical wounds and/or compromise of skin integrity.
* Individuals who cannot complete all phases of the study requirements.
* Individual requires use of an absorbent undergarment or catheter as the primary incontinence management strategy
* Individuals who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Miller, Study Director — Medline Industries
Locations (1):
- Rochester Clinical Research, Inc., Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants are combined in one arm for the analysis because the first two positions are the same for all participants.
Groups:
- All Participants: Each participant will be provided with the FitRight ® System for the duration of the study. The study products will be used to collect real-life measurement data in order to assess the FitRight® System.
Period: Overall Study
Arm/Group | All Participants
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 37
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 18
  Female | 38
  Other | 0
  Decline to Answer | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Sensor Detection
Description: Evaluate the FitRight System sensor's ability to detect when an adult brief has absorbed enough liquid (~90-360mL) normal saline via a simulated urinary void to trigger an alert to change the brief in the sitting, supine, and right or left side positions.
Time Frame: 5 minutes after each amount (90-360 milliliters) saline is poured into the brief. There could be up to four pours for each brief and 3 briefs (one for each position).
Population: Four participants were removed from the analysis because of deviations. The measure type mean was chosen below because the unit of measure is the percentage of passes.
Measure: Mean (95% Confidence Interval); unit: percentage of passes
Groups:
- All Participants: Each participant will be provided with the FitRight ® System for the duration of the study. The study products will be used to collect real-life measurement data in order to assess the FitRight® System.
  Wetness Sensing System Validation: Participants will use the Wetness Sensing System in a simulated setting in the sitting, supine and side position (participants are randomized to either the left or right side position).
Arm/Group | All Participants
Number analyzed (Participants) | 52
percentage of passes | 96.15 [0 to 100]

2. Secondary Outcome: Rewet Test
Description: Determine the FitRight Brief's residual volume capacity. In a subset of 22 participants, evaluate the FitRight Brief after the brief has absorbed the maximum amount of liquid normal saline via a simulated urinary void (360mL) in the sitting position and then weighed via the rewet procedure.
Time Frame: 10 minutes after the 360 milliliters saline is poured into the brief.
Population: A convenient subset of the first 22 completed participants was recruited. The unit of measure below is percent change in paper weight from dry.
  for the rewet procedure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | All Participants
Number analyzed (Participants) | 22
percent change | 18.73 (25.36)

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT05454813/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT05454813/ICF_001.pdf